CLINICAL TRIAL: NCT06574555
Title: Determination of the 90% Effective Dose of the Initial Bolus of Norepinephrine in Elective Cesarean Section: An Up-Down Study
Brief Title: Norepinephrine ED90 Bolus After Spinal Anesthesia in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Hector J. Lacassie, MD, Principal Investigator, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 240816002
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hypotension; Hypertension; Nausea; Pain; Arrhythmia
Keywords: Hypotension; Hypertension; Nausea; Pain; Arrhythmia
MeSH Terms: conditions — Hypotension; Hypertension; Nausea; Pain; Arrhythmias, Cardiac | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Experimental): Patients will be randomly assigned to sequence A who receive the study drug, norepinephrine. The initial bolus doses of norepinephrine will be 0.15 µg/kg.
  Interventions: Drug: Norepinephrine
- Sequence B (Experimental): Patients will be randomly assigned to sequence B who receive the study drug, norepinephrine. The initial bolus doses of norepinephrine will be 0.13 µg/kg.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — The outcome of patient n in each sequence will determine the dose to be allocated patient n+1.
  Successive doses will be determined with the up-and-down k-in-row design method for ED90 determination:
  * Failure: the dose should be increased in one level (+0.02 µg/kg) after failure to respond (arterial hypotension);
  * Success: decrease in one level (-0.02 µg/kg) upon successful response (no arterial hypotension), but only after observing at least k-consecutive positive responses at the same dose (in this case, k=7); otherwise, remain at the same dose.
  This will be done until each sequence completes n=30.

SUMMARY:
The investigators are aiming to determine what is the effective intravenous dose required of an initial bolus of norepinephrine prior to a maintenance infusion to prevent a 20% decrease in maternal blood pressure from baseline following the administration of spinal anesthesia for elective cesarean section in healthy parturients

DETAILED DESCRIPTION:
Previous studies have focused on determining the most appropriate doses for infusion administration of norepinephrine, and although current data allows us to conclude that the optimal initial dose would be around 0.05 mcg/kg/min, there are still reasonable doubts regarding the initial bolus dose prior to an infusion.

The primary outcome is to determine the 90% effective dose (ED90) of an initial bolus of norepinephrine in elective cesarean section under spinal anesthesia to prevent arterial hypotension.

The investigators hypothesize that the bolus ED90 of norepinephrine will be in the vicinity of 0.15 μg/kg, taking as reference the lower limit of a previous study (Lyu et. al.) and the dose used in equipotency studies with phenylephrine.

After approval by the Ethics Committee of Pontificia Universidad Católica de Chile and obtaining written informed consent, full-term pregnant patients, ASA II or III, scheduled for elective cesarean section will be prospectively included. The study will be registered in Clinical Trials and will be guided by the guidelines of the Helsinki declaration.

Inclusion criteria will be age between 18 and 40 years, elective caesarean section and singleton term pregnancy. Exclusion criteria will be hypertensive disorders of pregnancy; cardiovascular disease; baseline systolic BP <100 mmHg; height less than 145 cm or greater than 180 cm; weight less than 40 kg or greater than 100 kg, need for uterine exteriorization during surgery or coagulation disorders. The study will follow the 2010 Consolidated Standards for Reporting Trials (CONSORT) guidelines.

Patients will be randomly assigned to two sequences (A and B) who receive the study drug, norepinephrine. The initial bolus doses of norepinephrine will be 0.15 and 0.13 µg/kg.

Patients, the anesthesiologist involved in the patient's care, surgeons, data collectors and outcome adjudicators will be blinded to the initial dose of norepinephrine administered.

Anesthetic care will be according to institutional standards, which include preoperative fasting and non-invasive hemodynamic monitoring. After arrival in the operating room, patients will be positioned supine with left lateral tilt, to measure baseline blood pressure (BP) and heart rate after a brief resting period and averaging 3 consecutive measurements in which systolic BP varies <10%.

A peripheral intravenous (IV) line (caliber ≥18G) will be placed into an upper extremity vein under local anesthesia. Continuous low-rate fluids will be administered for patency purposes, but without prior hydration (pre-hydration). The patients will then be positioned in the left lateral decubitus position for the anesthetic puncture.

After skin disinfection and infiltration of the skin with 2% w/v lidocaine, subarachnoid anesthesia will be performed. A 25G Whitacre spinal needle (Pencan Braun, Germany) will be inserted through an introducer at the estimated intervertebral level L3-4 or L4-5. After confirming spontaneous cerebrospinal fluid reflux, 1.4 ml of hyperbaric bupivacaine 0.75% w/v (10.5 mg), fentanyl 0.4 ml (20 μg) and morphine 0.1 ml (50 μg) will be injected intrathecally. The patient will then be returned to the supine position with left lateral tilt for uterine displacement. Rapid intravenous cohydration will be started up to a total of 15 ml/kg, after which the infusion rate will be reduced to a maintenance rate. The upper sensory block level will be assessed using discrimination with ice. For comparison purposes, the upper dermatomal level of the blockade at 10 minutes after intrathecal injection will be recorded for each patient for warm discrimination and touch. The decision to allow surgery to commence will be based on the clinical judgment of the treating anesthesiologist.

Once the intrathecal anesthetic dose has been administered and the patient is positioned in the supine position, the study dose of norepinephrine will be administered as a rapid intravenous bolus. The first patients in each sequence receive a dose of 0.15 or 0.13 µg/kg (depending on the sequence they were randomised), the latter two levels lower than reported in a previous study in which the initial dose was calculated under these conditions9, which is recommended for this type of design11. This will be followed by a continuous infusion of norepinephrine at a dose of 0.05 µg/kg/min and titrating according to hemodynamic parameters.

The infusion syringe will contain 20 ml of norepinephrine solution (8 μg/ml) to be administered by a preprogrammed syringe pump at 0.05 µg/kg/min. The syringe for the initial bolus will be 20 ml and will contain norepinephrine at 1 µg/ml, allowing the dose corresponding to 0.13 or 0.15 µg/kg to be administered rounded to the nearest whole number (e.g. for 67 kg it is 10.05 µg, i.e. 10 ml (10 µg) will be administered).

Maternal blood pressure and heart rate will be recorded noninvasively every 1 minute immediately after spinal anesthesia until delivery, after which it will be monitored every 3 minutes.

The primary outcome will be the presence of arterial hypotension within 10 minutes of anesthesia administration. Post-spinal arterial hypotension will be defined as systolic BP decreasing to less than 80% of baseline. Norepinephrine (8 μg bolus) will be administered if the patient develops arterial hypotension despite study treatment. Severe post-spinal arterial hypotension will be defined if systolic BP decreases to <60% of baseline. Bradycardia will be defined as a heart rate below 50 beats per minute, where 0.3 mg of atropine will be administered. A rescue bolus will be re-administered if arterial hypotension or bradycardia is not corrected within one minute.

Arterial hypertension will be defined as a greater than 20% increase in baseline systolic BP and norepinephrine infusion will be discontinued.

Successive doses will be determined with the up-and-down k-in-row design method for ED90 determination:

* Failure: the dose should be increased in one level (+0.02 µg/kg) after failure to respond (arterial hypotension);
* Success: decrease in one level (-0.02 µg/kg) upon successful response (no arterial hypotension), but only after observing at least k-consecutive positive responses at the same dose (in this case, k=7); otherwise, remain at the same dose11.
* Reject: Any problem during the execution of the protocol that prevents the evaluation of the intervention (failure in spinal anesthesia, drug error, withdrawal from the study, etc.) will be considered as a reject, which will condition the administration of the same dose to the next patient randomized to that group.

The sequences will be run in parallel until the total sample size of each is reached.

Systolic BP and heart rate values will be recorded at the end of each BP measurement cycle. Oxygen will not be routinely administered. The attending anesthesiologist will be free to override the protocol and administer alternative or additional medications at any time if deemed clinically indicated based on his/her clinical judgment. This could include administration of additional bolus norepinephrine (8 µg), ephedrine (10 mg) or atropine (0.3 mg) intravenously for the treatment of bradycardia associated with arterial hypotension. Treatment of bradycardia not associated with arterial hypotension will be managed expectantly by discontinuing all study medications.

After fetal delivery and umbilical cord sample will be taken for blood gas and glycaemia. After placental separation a uterotonic will be administered according to standard institutional management.

Any manifestations secondary to the use of norepinephrine will be recorded, such as: headache, hypertension, pain on injection site or changes in skin colour. Nausea or vomiting during the study period shall also be recorded.

Cesarean delivery will be performed using a traditional Pfannenstiel technique, with no uterine exteriorization.

Statistical analysis The primary outcome of the study will be the incidence of arterial hypotension in the first 10 minutes after spinal anesthesia.

For the sample size calculation, a total of 60 patients will be considered, which is the general recommendation to be used to determine the 90% effective dose (ED90), which balances the minimum number of subjects and would still provide a useful estimate11. In addition, sample sizes N>40 will give an exact lower 95% confidence interval (95%CI) limit for probability of response of 0.76 for an estimate at ED90.

Data will be summarized descriptively using mean (standard difference (SD), median [interquartiles] and count (%) as appropriate. Gaussian distribution will be assessed using the D'Agostino Omnibus, Kolmogorov-Smirnov and normality plot methods.

The investigators will use the up-and-down k-in-a-row design method. The confidence intervals obtained can guarantee sufficient coverage for 95% in this type of design. We will estimate the 90% effective dose and 95% CI of norepinephrine to prevent arterial hypotension. The dose-response will be modelled using isotonic and probit regression, with and without the pooled adjacent violators algorithm (PAVA), as sensitivity analyses, in addition to the Firth penalised maximum likelihood estimation regression (Firth PMLE Regression). Probabilities of response (95%CI) will be estimated for all doses tested.

For secondary outcomes, comparisons will be made between groups and between patients with arterial hypotension versus those without, using Student t-, Mann-Whitney U- and Fisher exact statistics, as appropriate. Nominal data shall be compared using the χ2 test. A p-value<0.05 will be considered significant. Bonferroni and Tukey-Kramer corrections will be applied to keep the type I error (α) at 0.05 so that the significance criterion is p<0.017 (0.05/3) for blood pressure measurements that are repeated over time.

Statistical analyses will be performed in R (RStudio v. 2021.09.0 Build 351), jamovi ((https://www.jamovi.org), Stata 17.0, Stata Inc., College Station TX and Number Cruncher Statistical Systems (NCSS) 2024, NCSS Inc., Kaysville UT.

ELIGIBILITY:
Inclusion Criteria:

* Full-term singleton pregnant patients
* ASA II or III
* Scheduled for elective cesarean section
* Age between 18 and 40 years.

Exclusion Criteria:

* Hypertensive disorders of pregnancy
* Cardiovascular disease
* Baseline systolic BP <100 mmHg
* Height less than 145 cm or greater than 180 cm
* Weight less than 40 kg or greater than 100 kg
* Need for uterine exteriorization during surgery
* Coagulation disorders.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-02 (Actual)

PRIMARY OUTCOMES:
Hypotension | First 10 minutes after spinal anesthesia dose.
  The primary outcome will be the presence of arterial hypotension within 10 minutes of anesthesia administration. Post-spinal arterial hypotension will be defined as systolic BP decreasing to less than 80% of baseline.

SECONDARY OUTCOMES:
Maternal side effects | First 10 minutes after spinal injection
  Any manifestations secondary to the use of norepinephrine will be recorded, such as: headache, hypertension, pain on injection site or changes in skin colour. Nausea or vomiting during the study period shall also be recorded.
Fetal side effects | Until completion of the surgical procedure
  After fetal delivery and umbilical cord sample will be taken for blood gas and glycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Ivonne Vargas Celis, MD, Study Chair — Presidente, Comité Ético Científico Salud de la Universidad Católica
Locations (1):
- Hospital Clinico, Pontificia Universidad Catolica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
The whole database will be shared upon reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: november 2025-novembre 2027
Access Criteria: Researchers after reaonable request, looking at similar outcomes as ours.

REFERENCES:
- [Result] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Result] Ngan Kee WD, Khaw KS, Ng FF, Lee BB. Prophylactic phenylephrine infusion for preventing hypotension during spinal anesthesia for cesarean delivery. Anesth Analg. 2004 Mar;98(3):815-21, table of contents. doi: 10.1213/01.ane.0000099782.78002.30. PMID 14980943
- [Result] Ngan Kee WD, Lee SWY, Ng FF, Khaw KS. Prophylactic Norepinephrine Infusion for Preventing Hypotension During Spinal Anesthesia for Cesarean Delivery. Anesth Analg. 2018 Jun;126(6):1989-1994. doi: 10.1213/ANE.0000000000002243. PMID 28678073
- [Result] Ngan Kee WD, Khaw KS, Ng FF. Prevention of hypotension during spinal anesthesia for cesarean delivery: an effective technique using combination phenylephrine infusion and crystalloid cohydration. Anesthesiology. 2005 Oct;103(4):744-50. doi: 10.1097/00000542-200510000-00012. PMID 16192766
- [Result] Hasanin AM, Amin SM, Agiza NA, Elsayed MK, Refaat S, Hussein HA, Rouk TI, Alrahmany M, Elsayad ME, Elshafaei KA, Refaie A. Norepinephrine Infusion for Preventing Postspinal Anesthesia Hypotension during Cesarean Delivery: A Randomized Dose-finding Trial. Anesthesiology. 2019 Jan;130(1):55-62. doi: 10.1097/ALN.0000000000002483. PMID 30335625
- [Result] Chen Y, Guo L, Qin R, Xi N, Wang S, Ma Y, Ni X. Dose-Response Study of Norepinephrine Infusion for Maternal Hypotension in Preeclamptic Patients Undergoing Cesarean Delivery Under Spinal Anesthesia. Clin Pharmacokinet. 2024 Jun;63(6):847-856. doi: 10.1007/s40262-024-01381-4. Epub 2024 Jun 13. PMID 38869701
- [Result] Belin O, Casteres C, Alouini S, Le Pape M, Dupont A, Boulain T. Manually Controlled, Continuous Infusion of Phenylephrine or Norepinephrine for Maintenance of Blood Pressure and Cardiac Output During Spinal Anesthesia for Cesarean Delivery: A Double-Blinded Randomized Study. Anesth Analg. 2023 Mar 1;136(3):540-550. doi: 10.1213/ANE.0000000000006244. Epub 2022 Oct 24. PMID 36279409